CLINICAL TRIAL: NCT03320551
Title: Can A Nutrition Education Immersion Program Foster Sustainable Improvements in Clinical Parameters Over Time?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Whole Foods, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB201702439
Record Dates: First submitted 2017-10-18; First posted 2017-10-25 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Behavior
Keywords: Education
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition Education Immersion Program (Experimental): Assessing if a one week lifestyle interventions can lead to long term health benefits.
  Interventions: Behavioral: Immersion program

INTERVENTIONS:
Behavioral: Immersion program — Evaluate the impact of an already established one week long lifestyle immersion program sponsored by Whole Foods, Inc for their employees on anthropomorphic, clinical labs such as lipid levels, blood sugar and other markers of nutrition, quality of life and activity levels at baseline, at the end of the program and at 3 and 6 months

SUMMARY:
Nutrition and Education Immersion program sponsored by WholeFoods, Inc. for their employees.

DETAILED DESCRIPTION:
An ongoing Nutrition and Education Immersion program is currently ongoing that is supported by Whole Foods, Inc. for their employees. Eighty employees have previously agreed to attend a one week nutrition education and immersion program October 14-21, 2017. This program will involve nutrition education seminars, exercise and support classes that they are scheduled to attend. All meals are provided. They will all be 100% plant based with low oil. All employees will complete a dietary survey at the beginning of the study. Clinical parameters will be tested at start and end of the program. The majority of the lectures are CME certified by Rush University.

All participants will be approached for participation on day one to allow for the collection of the data being obtained as part of the existing project. In addition to the data from the program, this project will include a lab draw for nutritional markers at baseline and at the end of the immersion program, a dietary survey, SF-36, and DASI at baseline. Participants will be contacted by phone at months 3 and 6 and will be asked to complete the dietary survey, SF-36, and DASI. In addition, self-reported weight will be collected, and occurrence of health events (hospitalizations, new diagnoses). This will end their participation.

ELIGIBILITY:
Inclusion Criteria:

* 18yrs or older
* all comers with and without cardiovascular disease risk factors
* are attending the one week lifestyle immersion program sponsored by Whole Foods

Exclusion Criteria:

-unwilling to provide consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Weight | Up to 6 months
  Self Reported by participating subject

SECONDARY OUTCOMES:
Mediterranean Diet Survey | Up to 6 months
  Diet Survey which is a standardized survey used to access patient nutritional intake Minimum Score is 0 points and Maximum Score is 15 points
36 Item Short Form Survey | Up to 6 months
  SF-36 Quality of Life questionnaire which is a set of generic, coherent and easily administered quality of life measures.
Duke Activity Status Index | Up to 6 months
  DASI(Duke Activity Status Index) which is a 12 item questionnaire that utilizes self reported physical capacity to estimate peak metabolic equivalents and has been shown to be a valid measurement of functional capacity.
  Score is based on the sum of "yes" replies and a value is given.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Aggarwal, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health, Gainesville, Florida
  - Naples Beach Hotel and Golf Club, Naples, Florida

IPD SHARING:
Plan to Share IPD: No